CLINICAL TRIAL: NCT01481220
Title: A Pilot Phase I Dose Finding Safety Study of a Thrombopoietin-receptor Agonist, Eltrombopag, in Patients With Myelodysplastic Syndrome Treated With Azacitidine
Brief Title: Safety Study of Eltrombopag Combined With Azacitidine to Treat Myelodysplastic Syndrome (MDS)
Acronym: NMDSG10A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nordic MDS Group (Network)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-023663-18
Record Dates: First submitted 2011-11-17; First posted 2011-11-29 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Myelodysplastic Syndrome; Thrombocytopenia
Keywords: Myelodysplastic syndrome; azacitidine; Eltrombopag; Thrombopoietin-receptor agonist; Thrombocytopenia; Transfusion dependency; Safety study
MeSH Terms: conditions — Myelodysplastic Syndromes; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacitidine + Eltrombopag (Experimental)
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — In this study 4 different doses of oral eltrombopag (50mg, 100mg, 200mg and 300mg) will be tested. A modified 3+3 patient cohorts design will be used so no new patients are accepted to start on a higher dose without prior tolerance at the previous dose. Patients will be given eltrombopag once daily starting one week before the start of azacitidine treatment and then continue throughout the study, which duration will be approximately 3 months (three Azacytidine cycles). Patients will be evaluated continuously by clinical and laboratory assessments as well as bone marrow examinations during the treatment period until 4 weeks after discontinuation of Eltrombopag. Response, AEs/SAEs and DLTs will be monitored throughout the study.

SUMMARY:
Patients with Myelodysplastic Syndromes (MDS) often suffer from low platelet levels which may lead to bleeding complications. Treatment with cytotoxic agents can decrease the platelet levels further. Eltrombopag is a relatively new drug that increases the platelet level in the blood by working directly on the bone marrow. It is available for treatment of the disease Immunological Thrombocytopenic Purpura (ITP). In this study patients with MDS and low platelet levels that are treated with the cytotoxic agent Azacitidine will also receive Eltrombopag. The administration of Eltrombopag to MDS patients treated with Azacitidine may result in less dose reductions and less treatment delays for Azacitidine and may reduce the need for thrombocyte transfusions and lower the risk of bleeding complications.

This is a phase I study, meaning that our major goal is to investigate the safety and tolerability for Eltrombopag in this patient group. It will also generate a basis for a phase II-III-study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (18 years of age or older) with advanced MDS or sAML/MDS requiring treatment with Azacitidine as approved by EMEA:

   * MDS classified as Intermediate 2-risk or high risk according to the international prognostic scoring system (IPSS) or
   * Chronic myelomonocytic leukaemia (CMML) with 10-29% bone marrow blasts without myeloproliferative disease or
   * Acute myeloblastic leukaemia (AML) with 20-30% bone marrow blasts with multilineage dysplasia according to the WHO classification.
2. Platelet counts < 75 x 109 /L at start of Azacitidine treatment.
3. Subjects must have platelet count and platelet transfusion data available over a period of 4 weeks prior to inclusion.
4. During the 8 weeks prior to inclusion in study, subjects must have a baseline bone marrow examination including all of the following:

   * cytomorphology to confirm bone marrow blasts
   * cytogenetics
5. ECOG Status 0-2.
6. Subject is able to understand and comply with protocol requirements and instructions.
7. Subject has signed and dated informed consent.
8. Adequate baseline organ function defined by the criteria below:

   * total bilirubin (except for Gilbert's Syndrome) </= 1.5xULN
   * ALT and AST </= 3xULN
   * creatinine </= 2.5 xULN
9. Subject is practicing an acceptable method of contraception (documented in CRF).Female subjects (or female partners of male subjects) must either be of non childbearing potential (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or post-menopausal > 1 year), or of childbearing potential and use 1 of the following highly effective methods of contraception (i.e., Pearl Index < 1.0%) from 2 weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study:

   * Complete abstinence from intercourse;
   * Intrauterine device (IUD);
   * Two forms of barrier contraception (diaphragm plus spermicide, and for males condom plus spermicide);
   * Male partner is sterile prior to entry into the study and is the only partner of the female;
   * Systemic contraceptives (combined or progesterone only).

Exclusion criteria:

1. Subjects with a diagnosis of acute promyelocytic leukemia.
2. Patients with short life expectancy (less than 3 months)
3. Patients with bone marrow fibrosis that does not allow bone marrow aspiration (so-called "dry tap") or fibrosis grade II or III (grading according to European consensus on grading bone marrow fibrosis.
4. History of treatment for cancer other than MDS or sAML/MDS with systemic chemotherapy and/or radiotherapy within the last 2 years.
5. Patients with clinically significant splenomegaly, or > 16 cm spleen in length measured by ultrasound
6. Patients with known liver cirrhosis
7. Patients with East Asian ancestry such as Chinese, Japanese, Taiwanese or Korean.
8. History of treatment with romiplostim or other TPO-R agonists.
9. subjects with a QTc > 450 msec (QTc > 480 msec for subjects with Bundle Branch Block).
10. Subjects with known thrombophilic risk factors. Exception: Subjects for whom the potential benefits of participating in the study outweigh the potential risks of thromboembolic events, as determined by the investigator.
11. Female subjects who are nursing or pregnant (positive serum or urine Beta-human chorionic gonadotropin [B-hCG] pregnancy test) at screening or pre-dose on Day 1.
12. Current alcohol or drug abuse.
13. Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
14. Active and uncontrolled infections.
15. Subjects infected with Hepatitis B, C or Human Immunodeficiency Virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability parameters | week 26
  Including:
  * Non-hematological clinical, laboratory Grade 3/Grade 4 toxicities
  * Change in bone marrow or peripheral blood blast counts from baseline
  * Adverse events and interactions at increasing doses of eltrombopag

SECONDARY OUTCOMES:
Azacitidine treatment delays and dose reductions | week 26
Need for thrombocyte transfusions | week 26
Bleeding complications | week 26
Possible signs of antineoplastic effects (blood values and bone marrow picture) | week 26

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Svensson, M.D., Study Director — Nordic MDS Group
Locations (1):
- 4 Locations, Uppsala, Stockholm, Göteborg, Umeå, Sweden